CLINICAL TRIAL: NCT02195934
Title: The Orange Juice and Cardiovascular Disease Study
Acronym: OJ & CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: European Commission (Other); Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IFR03/2014; 14/EE/0219 (Other: NRES Committee East of England - Norfolk); 155431 (Other: NIHR Coordinated System for Gaining NHS permission (NIHR CSP)); 2014GP23 (Other: South Norfolk CCG)
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-04

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease, blood orange juice, anthocyanins
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard orange juice (OJ) followed by blood OJ (Other): This randomized 2-way cross over study will compare the effect of blood orange juice with that of a standard (blonde) orange juice consumed daily for 28 days, on markers of cardiovascular disease, with a 3 week washout period in between.
  Interventions: Other: Standard (blonde) orange juice; Other: Blood orange juice
- Blood orange juice followed by standard OJ (Other): This randomized 2-way cross over study will compare the effect of blood orange juice with that of a standard (blonde) orange juice consumed daily for 28 days, on markers of cardiovascular disease, with a 3 week washout period in between.
  Interventions: Other: Standard (blonde) orange juice; Other: Blood orange juice

INTERVENTIONS:
Other: Standard (blonde) orange juice — Consumption of 500ml standard (blonde) orange juice daily for 28 days
Other: Blood orange juice — Consumption of 500ml blood orange juice daily for 28 days

SUMMARY:
This study aims to compare the effect of an anthocyanin-rich blood orange juice with a standard (no anthocyanin) blonde orange juice on markers of cardiovascular disease (CVD).

Participants aged between 25 and 84 years of age will be recruited into a single arm, two way cross-over study based on their waist measurement, with 42 individuals required to complete the study. Participants will each receive two interventions in a randomised order: 500mL blood orange juice daily for 28 days, and 500ml standard (blonde) orange juice daily for 28 days.

Prior to each intervention there will be a 2 week "run in period" where participants will be asked to avoid consuming foods rich in anthocyanins. After the first 28 day intervention period, there will be a 3 week wash out period after which the participants will be asked to then drink the other juice for 28 days. The 500 mL of blood orange juice contains approximately 50mg of anthocyanins, whereas the standard juice contains none.

Blood samples will be collected for the preparation of plasma and peripheral blood mononuclear cells (PBMCs) for the analysis of anthocyanin metabolite concentrations, transcriptomics and CVD risk markers. Urine samples will be collected and urinary excretion of anthocyanin metabolites will be quantified. Other measurements will include pulse wave analysis, pulse wave velocity, central blood pressure, waist and hip circumference, blood glucose, glycated haemoglobin (HbA1C) and insulin concentrations, and various measurements using the TANITA machine which include weight, fat mass, muscle mass, fat percentage, fat-free mass, total body water, bone mass, metabolic age, basal metabolic rate, visceral fat rating, and degree of obesity. All measurements and samples will be taken at baseline and post intervention for each phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 25-84 years
* Waist measurement

  * Caucasians: Men > 102cm (40inches); Women >88cm (34inches)
  * Asians: Men> 90cm (35inches); Women 80cm (31inches)

Exclusion Criteria:

* Those unable to give written informed consent
* Those unwilling to provide general practitioner (GP) details
* Regular prescribed medication that may affect study outcome. This will be assessed on an individual basis-not including statins
* Over-the-counter (non-prescribed) medication that may affect the study data. This will be assessed on an individual basis.
* Allergy to the test juice drink or the actual fruit itself
* Chronic medical conditions requiring active treatment. This will be assessed on an individual basis
* Those already consuming blood orange juice, unless they are willing to discontinue consumption for 2 weeks prior to starting the study.
* Diagnosed diabetics;
* Peri-menopausal women (defined as: when there is a permanent change in menstrual cycle)
* Women on hormone replacement therapy (HRT) for less than one year
* On thyroxine for less than one year
* Women who are pregnant, have been pregnant within the last 12 months or who are breastfeeding
* Those taking aspirin (prescribed or self-prescribed)
* All blood pressure medication
* Those individuals who happen to be on statins will be excluded if they have been on statins for less than 3 months; or if they are not taking on a daily basis; or those who have recently changed their dosage of statins. This will be assessed on an individual basis
* Those on regular medication for hypercoagulation and inflammatory conditions e.g. corticosteroids and asthma. The intermittent use of an inhaler will be discussed on an individual basis
* Those who have had a cardiovascular event such as stroke, myocardial infarction (heart attack) or trans ischemic attacks in the past and deemed unsuitable for participation in the study. This will be discussed with the medical adviser on an individual basis
* Peripheral vascular disease including claudication
* Consumption of fish oil supplements (unless participant is willing to discontinue their use 8 weeks prior to the start of the intervention- all other supplements will be assessed on an individual basis
* Parallel participation in another research project which has involved dietary intervention and/or sampling of blood
* Any person related to or living with any member of the study team
* Participation in another research project which involves blood sampling within the last four months unless the total blood from both studies (including this one) does not exceed 470mL)
* Those who have donated or intend to donate blood within 16 weeks of the first and last study samples
* Gastrointestinal disease (excluding hiatus hernia) unless symptomatic or study intervention/procedure is contraindicated
* Those undergoing any on-going clinical investigations with their GP or hospital clinic.
* Those who have had throat surgery or neck injury
* Those with internal medical devices

Screening exclusion criteria

* Results of the eligibility screening that indicate or are judged by the Institute of Food Research Human Nutrition Unit (HNU) medical adviser to be indicative of a health problem which could compromise the well-being of the participant if they participated or could affect the study data.
* BMI <19.5
* Weight >180kg (28stones)
* Fasting total cholesterol > 8.0mmol/L
* Haemoglobin Men <13.8g/dL (8.56mmol/L) Women <12.1g/dL (<5.51mmol/L)
* Fasting glucose >6mmol/L
* Blood pressure <90/50mmHg or 95/55mmHg if symptomatic; >160/100mmHg
* Anyone with any internal medical devices (incompatible with the TANITA)

Ages: 25 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 28 days (4 weeks)
  The primary outcome measure will be the change in concentration of LDL cholesterol as a result of the daily consumption of standard (blonde) orange juice or blood orange juice for 28 days (4 weeks).

SECONDARY OUTCOMES:
CVD biomarkers | 28 days (4 weeks)
  The secondary outcome measure include measuring the change in concentration of levels of other markers of CVD, HDL, total cholesterol, nitrites, nitrates, nitrosols, interleukin 6, high sensitivity C reactive protein, Dglucose, insulin and endothelin 1 as a result of daily consumption of standard (blonde) orange juice or blood orange juice for 28 days (4 weeks).

OTHER OUTCOMES:
Gene expression | 28 days (4 weeks)
  The assessment of the activity of genes (gene expression) as a result of the daily consumption of standard (blonde) orange juice and blood orange juice for 28 days (4 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Kroon, PhD, Study Director — Quadram Institute Bioscience; Charlotte N Armah, PhD, Principal Investigator — Quadram Institute Bioscience; Joanne F Doleman, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Hollands WJ, Armah CN, Doleman JF, Perez-Moral N, Winterbone MS, Kroon PA. 4-Week consumption of anthocyanin-rich blood orange juice does not affect LDL-cholesterol or other biomarkers of CVD risk and glycaemia compared with standard orange juice: a randomised controlled trial. Br J Nutr. 2018 Feb;119(4):415-421. doi: 10.1017/S0007114517003865. PMID 29498348